CLINICAL TRIAL: NCT04530032
Title: Ketogenic Diet & Functional Recovery in Moderate to Severe Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Brenda Bartnik Olson, PhD, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5200137
Record Dates: First submitted 2020-08-11; First posted 2020-08-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; ketogenic diet; metabolism; spectroscopy; cerebral blood flow; modified Atkins diet
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBI KD/MAD (Experimental): TBI subjects on a ketogenic/modified Atkins diet
  Interventions: Other: ketogenic/modified Atkins diet
- TBI SD (Sham Comparator): TBI subjects on a standard (normal) diet
  Interventions: Other: Standard diet

INTERVENTIONS:
Other: ketogenic/modified Atkins diet — ketogenic/modified Atkins diet use
  Arms: TBI KD/MAD
Other: Standard diet — standard (normal) diet use
  Arms: TBI SD

SUMMARY:
Traumatic Brain Injury (TBI) represents a significant public health risk in the United States leaving many survivors with significant long term cognitive deficits and at risk for neurodegenerative diseases. Despite extensive research there are no pharmacological therapies which have demonstrated significant improvement in neurological or cognitive recovery. Changes in glucose metabolism are considered the hallmark metabolic response to TBI and ketosis has been proposed as a therapy to ameliorate metabolic dysfunction. This trial investigates the therapeutic potential of a ketogenic or modified Atkins diet on neurocognitive outcome following moderate-severe TBI.

DETAILED DESCRIPTION:
Traumatic Brain Injury (TBI) represents a significant public health risk in the United States leaving many survivors with significant long term cognitive deficits and at risk for neurodegenerative diseases. Despite extensive research there are no pharmacological therapies which have demonstrated significant improvement in neurological or cognitive recovery. Changes in glucose metabolism are considered the hallmark metabolic response to TBI and ketosis has been proposed as a therapy to ameliorate metabolic dysfunction. Further research is necessary to address the outstanding questions regarding outcome, dose, timing, route and duration of ketogenic diet (KD) or modified Atkins diet (MAD) therapy in clinical TBI. Using a multiparametric MRI and MR spectroscopy approach in conjunction with standardized neurological and neuropsychological assessments of outcome, disability, cognition, and quality of life, this trial will investigate the therapeutic potential of KD/MAD on 12 month outcome following moderate-severe TBI patients.

The purpose of this project is to:

1. Determine the effect of KD/MAD on cognitive and neurological outcome following moderate - severe TBI. To date clinical studies of ketone metabolism in TBI are severely limited and have focused primarily on ketometabolism and its effects on glucose metabolism without assessing functional or cognitive outcomes. This project directly assesses the effect of KD/MAD on measures of disability, attention, memory, processing speed, language, and executive function during ketosis and will determine whether its effects outlast the duration of the diet.
2. Identify the effects of KD/MAD on cerebral metabolism following moderate - severe TBI. While the use of ketogenic fuels is receiving greater attention, little is known about the effect of the KD/MAD on neuronal metabolism. This project will use MR spectroscopy to non-invasively measure NAA, a marker of neuronal metabolism during ketosis and outside the treatment window, which will deepen our understanding of the neuroprotective mechanisms of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* complicated mild (GCS 13-15), moderate (GCS 9 - 12) to severe (GCS ≤ 8) traumatic brain injury (TBI) between 2-30 days post injury
* Admitted to Loma Linda University surgical intensive care unit (SICU)

Exclusion Criteria:

* history of comorbid ischemic stroke following qualifying TBI
* history of premorbid brain injury with associated loss of consciousness
* history of psychiatric disorder
* history of premorbid neurological disorder or neurosurgical intervention
* pregnancy
* depressed GCS score due to acute intoxication
* liver dysfunction as defined by liver enzymes 5 times the upper limit of normal or chronic cirrhosis
* acute renal failure according to the Risk, Injury, Failure, Loss of kidney function, and End-stage kidenty disease (RIFLE) classification
* abdominal surgery during the same admission
* type 1 diabetes
* gastroparesis
* dyslipidemia
* severe asphasia
* known history of metabolic disorders that are a contradiction for ketogenic diet (KD) such as primary carnitine deficient, carnitine palmitoyltransferase (CPT) I or II deficiency, carnitine translocase deficiency, beta-oxidation defects, pyruvate carboxylase deficiency, or porphyria
* prealbumin (transthyretin) levels of <10 mg/dL within 3 days of admission
* Metal, implanted device (ICP monitor), pregnancy, claustrophobia, or other contraindication to MRI

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Neurological outcome | day 0 to 12 months
  The Disability Rating Scale (DRS) will be used to measure general functional changes as a result of the dietary intervention over a 6 month recovery period. This scale ranges from 0 (without disability) to a maximum score of 29 (extreme vegetative state).
Change in cerebral metabolism | day 0 to 12 months
  Single voxel magnetic resonance spectroscopy will be used to assess changes in cerebral metabolism as a result of the dietary intervention.

SECONDARY OUTCOMES:
Neurocognitive outcome: Trail Making Test, Part B | day 0 to 12 months
  A change in visual motor and visual spatial ability and mental flexibility as a result of the dietary intervention will be assessed over a 6 month period. Results are reported as the number of seconds required to complete the task with higher scores reveal greater impairment.
Neurocognitive outcome: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | day 0 to 12 months
  A change in cognitive improvement as a result of the dietary intervention will be assessed across 5 domains using the RBANS:
  Immediate Memory - List learning and Story Memory Visuospacial/Constructional - Figure Copy and Line Orientation Language - Picture naming and Semantic Fluency Attention - Digit Span and Coding Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall The five domain scores are combined as a total scale score. According to the RBANS manual, the possible values for the RBANS scores at the item, domain, and scale level are 0 to 89, 40 to 154, and 40 to 160.
Neurocognitive outcome: Delis Kaplan Executive Function System (D-KEFS) | day 0 to 12 months
  A change in executive function as a result of the dietary intervention will be assessed over a 6 month period using the verbal fluency and color word interference subtests of the D-KEFS. Achievement scores (total correct responses and total switching accuracy) will be measured using the D-KEFS Scoring Assistant software.
Neurocognitive outcome: 36 Item Short Form Survey (SF-26) | day 0 to 12 months
  Changes in quality of life as a result of the dietary intervention will be assessed over a 6 month period using the SF-36. Items are scored so that a high score defines a more favorable health state, with each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Bartnik-Olson, PhD, Principal Investigator — Loma LInda University Medical Center; Duc Tran, MD, Principal Investigator — Loma LInda University Medical Center
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No